CLINICAL TRIAL: NCT01961596
Title: Does Have a Short-term "Cooling Ice Spray" Application at the Lateral Ankle an Influence on the Time to Stability After a Forward Jump?
Brief Title: The Influence of a "Cooling Ice Spray " Application on the Time to Stability After a Forward Jump?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swanenburg (Other)
Responsible Party: Sponsor-Investigator, Swanenburg, PhD, Balgrist University Hospital
Organization: Balgrist University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: Balgrist 2013-0359; KEK-ZH-Nr. 2013-0359 (Other: Ethics commission of the Canton Zurich, Switzerland)
Record Dates: First submitted 2013-10-08; First posted 2013-10-11 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Healthy
Keywords: Cooling ice spray; Time to stability; Jump
MeSH Terms: interventions — Water

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- cooling ice (Experimental): A bursts of the "Cooling Ice Spray" over a period of 10 seconds (15 cm distance) will be applied at the dominant foot in before each test.
  After 2 days the measurements will be repeated with the other application.
  Interventions: Other: Cooling Ice Spray
- water (Placebo Comparator): A bursts of the water spray (room temperature over a period of 10 seconds (15 cm distance) will be applied at the dominant foot in before each test.
  After 2 days the measurements will be repeated with the other application.
  Interventions: Other: water

INTERVENTIONS:
Other: Cooling Ice Spray — A bursts of the "Cooling Ice Spray" over a period of 10 seconds (15 cm distance) will be applied at the dominant foot in before each test.
  Other Names: Perskindol Cool Spray
  Arms: cooling ice
Other: water — A bursts of the water spray (room temperature over a period of 10 seconds (15 cm distance) will be applied at the dominant foot in before each test.
  Other Names: Placebo water
  Arms: water

SUMMARY:
The aim of this study is to investigate the influence of a brief application of cold (by means of Cooling Ice Spray on the lateral ankle)on the time to stabilization of healthy subjects.

DETAILED DESCRIPTION:
In sports are "Cooling Ice Spray" applications after an injuries one of the most common and popular methods used. It is very popular mainly because of its analgesic effect and easy application. It is assumed that such application will not affect the athletes. Nevertheless after an application of cold a reduced nerve conduction velocity was measured, resulting in a reduction in pain and a reduced transmission rate. Usually the static equilibrium or the perception of joint position was investigated and not the time to stability. As far as we have been known so far been no study that has examined the impact of a brief application of cooling ice spray on the time to stability after dynamic function. Therefore this study what's to investigate the influence of "Cooling Ice Spray" on the time to stability after a forward jump.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults
* 18-45 age
* >3 Score "Tegner-Activity-Scale"

Exclusion Criteria:

* Cognitive deficits
* Physical disability
* Pain
* Injuries in the previous 6 weeks
* Non healed injuries at the leg
* Allergic reaction from cooling ice pray

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2013-10; Primary Completion 2014-02 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Time to stability | All measurements will be executed within 1hour. After 2 days the measurements will be repeated
  Immediately after the application the time to stability after a forward jump will be assessed.

SECONDARY OUTCOMES:
Skin temperature | All measurements will be executed within 1hour. After 2 days the measurements will be repeated
  Immediately after the application the Skin temperature will be assessed.
Side step time to stability | All measurements will be executed within 1hour. After 2 days the measurements will be repeated
  Immediately after the application the time to stability after side step will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Jaap Swanenburg, PhD, Principal Investigator — Balgrist Univeresty Hospital
Locations (1):
- Balgrist Univeresty Hospital, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No